CLINICAL TRIAL: NCT07343401
Title: Impact of Immunosuppressive Therapy of Sarcoidosis on Lymphoma Development
Brief Title: Sarcoidosis Immunotsuppressive Therapy and Lymphoma Development
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Sabry, lecturer, Alexandria University
Other Study IDs: Alexandria U; Alexandria University (Other: alex main university hospital)
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Sarcoidosis Lung
Keywords: lymphoma; sarcoidosis
MeSH Terms: conditions — Sarcoidosis, Pulmonary; Lymphoma; Sarcoidosis | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inclusion criteria include adult patients (≥16 years) with histologically confirmed sarcoidosis, rec: This is a prospective observational cohort study to be conducted in the Chest Diseases Department, Alexandria Main University Hospital. A total of 40 adult patients (≥16 years) with biopsy-proven sarcoidosis will be consecutively recruited between December 2024 and December 2025. All patients will be either newly starting or continuing immunosuppressive therapy for sarcoidosis.
  Interventions: Procedure: lymph node biopsy

INTERVENTIONS:
Procedure: lymph node biopsy — sarcoidosis diagnosis by lymph node biopsy excisiona or bronchoscopic

SUMMARY:
Impact of Immunosuppressive Therapy for Sarcoidosis on Lymphoma Development

DETAILED DESCRIPTION:
This is a prospective observational cohort study to be conducted in the Chest Diseases Department, Alexandria Main University Hospital. A total of 40 adult patients (≥16 years) with biopsy-proven sarcoidosis will be consecutively recruited between December 2024 and December 2025. All patients will be either newly starting or continuing immunosuppressive therapy for sarcoidosis. The treatment regimen-systemic corticosteroids, conventional steroid-sparing agents (methotrexate, azathioprine, or mycophenolate), or biologics (anti-TNF agents)-will be recorded but not altered by study design. Each patient will be followed prospectively for 12 months from enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria include adult patients (≥18 years) with histologically confirmed sarcoidosis, receiving or planned to receive immunosuppressive therapy

Exclusion Criteria:Patients with a prior history of lymphoma or other active malignancy, HIV infection, or other primary immunodeficiency will be excluded.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Prospective cohort
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be incident, biopsy-proven lymphoma during the 12-month follow-up. | 12 MONTHS
  LYMPH NODE BIOPSY EITHER EXCISIONAL OR BRONCHOSCOPIC
lymphoma development | 12 months
  lymph node biopsy excisional or bronchoscopic

CONTACTS AND LOCATIONS:
Overall Officials: ahmed mahmoud fawzy, professor, Principal Investigator — Alexandria University
Locations (1):
- Alexandria main university hospital, Alexandria, Asafra, Egypt

IPD SHARING:
Plan to Share IPD: No
not allowed in our department

REFERENCES:
- See also: pubmed — https://pubmed.ncbi.nlm.nih.gov/20594135/
- See also: national library of diseases — https://pubmed.ncbi.nlm.nih.gov/20594135/
- Available data/document: Statistical Analysis Plan: statistics — https://pubmed.ncbi.nlm.nih.gov/20594135/ — pending